CLINICAL TRIAL: NCT01719055
Title: A Global Prospective Observational Post-Market Study to Evaluate Long-Term Effectiveness of Neurostimulation Therapy for Pain
Brief Title: RELIEF - A Global Prospective Observational Post-Market Study to Evaluate Long-Term Effectiveness of Neurostimulation Therapy for Pain
Acronym: RELIEF
Status: Recruiting | Type: Observational
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: A7007; 90876777 (Other: BSC protocol number)
Record Dates: First submitted 2012-10-30; First posted 2012-11-01 (Estimated); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Pain
Keywords: stimulation; implantable; pulse generator; back pain; chronic pain; leg pain
MeSH Terms: conditions — Pain; Back Pain; Chronic Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Boston Scientific SCS Systems: Subjects permanently implanted with a Boston Scientific neurostimulation systems
  Interventions: Device: neurostimulation system

INTERVENTIONS:
Device: neurostimulation system — Trial stimulation period, followed by permanent implant of a neurostimulation system for subjects with a positive trial outcome

SUMMARY:
To compile characteristics of real-world clinical outcomes for Boston Scientific commercially approved neurostimulation systems for pain in routine clinical practice, when used according to the applicable Instructions for Use

- and -

To evaluate the economic value and technical performance of Boston Scientific commercially approved neurostimulation systems for pain in routine clinical practice

DETAILED DESCRIPTION:
The study is a prospective, multi-center, global, post-market study of Boston Scientific neurostimulation systems for pain.

The study treatment will consist of neurostimulation trial therapy with any commercially approved Boston Scientific Corporation neurostimulator for pain. Positive trials, subjects with a successful trial outcome, may progress to permanent implant of a neurostimulation system. Individualization of neurostimulation therapy for pain will be determined according to investigator discretion and site routine care, and in accordance with inclusion and exclusion criteria.

ELIGIBILITY:
Key Inclusion Criteria:

* Study candidate is scheduled to be trialed, on-label, with a commercially approved Boston Scientific neurostimulation system for pain, per local directions for use
* Signed a valid, IRB/EC-approved informed consent form
* 18 years of age or older

Key Exclusion Criteria:

* Contraindicated for Boston Scientific neurostimulation system
* Currently diagnosed with cognitive impairment, or exhibits any characteristic, that would limit study candidate's ability to assess pain relief or to complete study assessments

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects who exhibit an on-label indication for neurostimulation to relieve chronic intractable pain, according to the Instructions for Use, as applicable in each country or region
Sampling Method: Probability Sample
Enrollment: 4800 (Estimated)
Dates: Start 2012-11-19 (Actual); Primary Completion 2035-05 (Estimated); Study Completion 2035-05 (Estimated)

OTHER OUTCOMES:
Percent Pain Relief | Up to 60 months follow up
  Percent pain relief of targeted pain at 6, 12, 24, 36, 48, and 60 months follow up
Percent Pain Relief | Up to 60 months follow up
  Percent pain relief of low back pain at 6, 12, 24, 36, 48, and 60 months follow up
Percent Pain Relief | Up to 60 months follow up
  Percent pain relief of leg pain at 6, 12, 24, 36, 48, and 60 months follow up
Change in QoL | Up to 60 months follow up
  Change in quality of life as reported by the Subject at

CONTACTS AND LOCATIONS:
Overall Officials: Natalie Bloom Lyons, Study Director — Boston Scientific Corporation
Locations (116):
- United States (67):
  - Physicians Research Group, LLC, Phoenix, Arizona
  - Hope Research Institute, Phoenix, Arizona
  - Banner University Medical Center, Tucson, Arizona
  - Comprehensive Pain Management Center, Campbell, California
  - Coastal Research Institute, Carlsbad, California
  - Pain Medicine Associates, Inc., Fountain Valley, California
  - Metropolitan Pain Management Consultants Inc., Sacramento, California
  - Huntley Pain Specialists, San Diego, California
  - Conejo Pain Specialists, Thousand Oaks, California
  - Denver Back Pain Specialists, Greenwood Village, Colorado
  - Orlando Health Neuroscience Institute, Inc, Clermont, Florida
  - South Lake Pain Institute, Inc, Clermont, Florida
  - University of Florida Shands Hospital, Gainesville, Florida
  - Louis J. Raso, MD, PA, Jupiter, Florida
  - Advanced Interventional Pain Management and Research Clinic, Inc., Miami Gardens, Florida
  - JM Clinical Research, South Miami, Florida
  - Tallahassee Neurological Clinic, PA, Tallahassee, Florida
  - Orthopedic Research Foundation, Savannah, Georgia
  - Pain Care, LLC, Stockbridge, Georgia
  - Northwestern Memorial Hospital - Neurosurgery Outpatient Clinic, Chicago, Illinois
  - Chicago Anesthesia Pain Specialists, Chicago, Illinois
  - Global Scientific Innovations - Advanced Pain Care Clinic, Evansville, Indiana
  - Summit Research Institute, Fort Wayne, Indiana
  - Goodman Campbell Brain and Spine, Greenwood, Indiana
  - American Health Network of Indiana, LLC, Muncie, Indiana
  - Research Medical Center, Lenexa, Kansas
  - Neuroscience Associates of Northern Kentucky, Crestview Hills, Kentucky
  - Bux Pain Management, Danville, Kentucky
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - Willis-Knighton River Cities Clinical Research Center, Shreveport, Louisiana
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Brookline, Massachusetts
  - Michigan Pain Specialists, Ann Arbor, Michigan
  - Insight Institute of Neurosurgery & Neuroscience, Flint, Michigan
  - Forest Health Medical Center, Ypsilanti, Michigan
  - Jackson Anesthesia Pain Center, LLC, Jackson, Mississippi
  - Midwest Pain Center, Chesterfield, Missouri
  - Saint Louis Pain Consultants, Chesterfield, Missouri
  - KC Pain Centers, Lee's Summit, Missouri
  - Hope Research Institute, Las Vegas, Nevada
  - Albany Medical Center, Albany, New York
  - New York Presbyterian Hospital, New York, New York
  - University of Rochester, Rochester, New York
  - Montefiore Medical Center, The Bronx, New York
  - Spine and Skeletal Pain Medicine, Utica, New York
  - Carolinas Research Institute, PLLC, Huntersville, North Carolina
  - Raleigh Neurology Associates, P.A., Raleigh, North Carolina
  - The Center for Clinical Research, LLC, Winston-Salem, North Carolina
  - Case Western Reserve University, Cleveland, Ohio
  - Ohio State University Medical Center, Columbus, Ohio
  - University of Toledo Medical Center, Toledo, Ohio
  - Pacific Sports and Spine, LLC, Eugene, Oregon
  - Fox Chase Pain Management, Trevose, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Florence Neurosurgery and Spine, Florence, South Carolina
  - PCPMG Clinical Research Unit, LLC, Greenville, South Carolina
  - Channel Research, Pawleys Island, South Carolina
  - Balcones Pain Consultants, Austin, Texas
  - Institute of Precision Pain Medicine, Corpus Christi, Texas
  - Spine Works Institute, North Richland Hills, Texas
  - Spine Team Texas, Rockwall, Texas
  - Precision Spine Care, Tyler, Texas
  - Washington Center for Pain Management, Bellevue, Washington
  - EvergreenHealth Pain Care, Kirkland, Washington
  - Swedish Neuroscience Institute, Seattle, Washington
  - West Virginia University Hospitals, Morgantown, West Virginia
  - Advanced Pain Management Appleton, Greenfield, Wisconsin
- CENIT Centro de Neurociencias, Investigacion y Tratamiento, Buenos Aires, Argentina
- Australia (8):
  - Interventus Pain Specialists, Auchenflower
  - Hunter Clinical Research, Broadmeadow
  - Hunter Pain Clinic, Broadmeadow
  - Green Lizard Science, Claremont
  - Sydney Spine and Pain Pty Ltd, Hurstville
  - Sunshine Coast Clinical Research, Noosa
  - Pain Matrix, Waurn Ponds
  - Pain Medicine of South Australia, Wayville
- Belgium (2):
  - AZ Sint-Lucas, Ghent
  - AZ Delta, Roeselare
- Canada (3):
  - London Health Sciences Centre, London
  - Hopital de Enfant-Jesus, Québec
  - Regina General Hospital, Regina
- Colombia (2):
  - Fundacion Clinica Valle del Lili, Cali
  - Fundacion Cardiovascular de Colombia Floridablanca, Floridablanca
- Odense University Hospital, Odense, Denmark
- Germany (5):
  - Universitatsklinik Charite Berlin, Berlin
  - University KH Bonn, Bonn
  - Uniklinik Köln, Cologne
  - Universitaetsklinikum Dusseldorf, Düsseldorf
  - Algesiologikum, München
- Israel (2):
  - Sheba Medical Center, Ramat Gan
  - Tel Aviv Sourasky Medical Center, Tel Aviv
- Italy (2):
  - Fondazione Salvatore Maugeri IRCCS, Pavia
  - Azienda Ospedaliero Universitaria Pisana, Pisa
- Japan (4):
  - Kobe University Hospital, Kobe
  - Hyogo College of Medicine Hospital, Nishinomiya-shi
  - Okayama University Hospital, Okayama
  - Sakai Hospital Kinki University Faculty of Medicine, Sakaishi
- Ziekenhuis Rijnstate, Velp, Netherlands
- Spain (10):
  - Hospital General de Ciudad Real, Ciudad Real
  - Hospital La Paz, Madrid
  - Hospital La Princesa, Madrid
  - Hospital Puerta de Hierro, Madrid
  - Hospital Universitario Infanta Elena, Madrid
  - Clinica Universidad de Navarra, Pamplona
  - Hospital Donostia, San Sebastián
  - H. Marques De Valdecilla, Santander
  - Hospital Virgen De La Salud, Toledo
  - Hospital General de Valencia, Valencia
- Sahlgrenska University Hospital, Gothenburg, Sweden
- Ospedale Regionale di Lugano, Viganello, Switzerland
- United Kingdom (6):
  - Basildon and Thurrock University Hospitals NHS, Basildon
  - Southmead Hospital Bristol, Bristol
  - The General Infirmary, Leeds
  - Chelsea and Westminster Hospital, London
  - St. Bartholomews Hospital, London
  - Royal National Orthopaedic Hospital, Stanmore

REFERENCES:
- [Derived] Rauck RL, Loudermilk E, Thomson SJ, Paz-Solis JF, Bojrab L, Noles J, Vesper J, Atallah J, Roth D, Hegarty J, Prud'Homme M, Phillips GM, Smith SG, Ibrahim M, Willoughby CD, Obray JB, Gupta M, Paez J, Berg AP, Harrison NJ, Maino P, Mambalam P, McCarty M, Towlerton G, Love-Jones S, Ahmed S, Lee A, Shah B, Goor-Aryeh I, Russo MA, Varela N, Phelps JB, Cid J, Fernandez T, Perez-Hernandez C, Keehn D, Rosenow JM, Haider N, Parrent AG, Lawrence MM, Georgius P, Demartini L, Mendiola A, Mehta V, Thoma R, Israel AF, Carolis G, Bhatia S, Green M, Villarreal A, Crooks MT, Gwinn RP, Pilitsis JG, Sato H, Vega SM, Hillegass MG, Carnes P, Scherer C, Brill S, Yu J, Brennan JJ, Gatzinsky K, Navani A, Snook LT Jr, Bujedo BM, Andres Ares J, Murillo A, Trobridge AT, Assil K, Shah J, McLeod C, Buwembo J, Coster O, Miller N, Sanapati M, Mikhael M, Przkora R, Sukenaga N, Raso LJ, Calodney AK, Caceres Jerez LE, Uchiyama T, Kallewaard JW, Chandler B, Piedimonte F, Candido KD, Weaver TE, Agari T, Holthouse D, Woon R, Patel N, Lechleiter K, Jain R. Long-term safety of spinal cord stimulation systems in a prospective, global registry of patients with chronic pain. Pain Manag. 2023 Feb;13(2):115-127. doi: 10.2217/pmt-2022-0091. Epub 2023 Jan 24. PMID 36691862